CLINICAL TRIAL: NCT03687736
Title: A Multicenter, Open-Label, Interventional Study to Evaluate Subject Satisfaction of AbobutulinumtoxinA Treatments in Moderate to Severe Glabellar Lines
Brief Title: Subject Satisfaction With AbobutulinumtoxinA Treatment
Acronym: DREAM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 43USD1802
Record Dates: First submitted 2018-09-19; First posted 2018-09-27 (Actual); Results first posted 2020-03-18 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2020-03

CONDITIONS: Glabellar Frown Lines
MeSH Terms: interventions — abobotulinumtoxinA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- AbobotulinumtoxinA (Other): Open-label
  Interventions: Biological: AbobotulinumtoxinA

INTERVENTIONS:
Biological: AbobotulinumtoxinA — AbobotulinumtoxinA treatment in the glabellar region at Baseline and Month 6

SUMMARY:
An interventional Phase 4 study to assess subject satisfaction with abobotulinumtoxinA treatment.

DETAILED DESCRIPTION:
Following signature of informed consent and the screening process, eligible subjects were treated at the Baseline visit (Day 0) with abobotulinumtoxinA in the glabellar region. Subjects were re-treated at the Month 6 visit.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to Severe Glabellar Lines at Maximum Frown
* Understands study requirements and signs an informed consent

Exclusion Criteria:

* Known allergy to any component of study product
* Pregnant or breast feeding or intending to get pregnant during the study
* Botulinum toxin treatment in the face within 9 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2019-11-07 (Actual); Study Completion 2019-12-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Galderma Study Site, Los Angeles, California
  - Galderma Study Site, San Francisco, California
  - Galderma Study Site, Santa Monica, California
  - Galderma Study Site, Greenwood Village, Colorado
  - Galderma Study Site, Chicago, Illinois
  - Galderma Study Site, Omaha, Nebraska

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- abobotulinumtoxinA: open-label
  AbobotulinumtoxinA: AbobotulinumtoxinA treatment in the glabellar region
Period: Overall Study
Arm/Group | abobotulinumtoxinA
Started | 120
Completed | 110
Not Completed | 10
Not completed — Lost to Follow-up | 7
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | AbobotulinumtoxinA
Number analyzed (Participants) | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 120
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 109
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 107
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 120
Toxin Naive Status [Count of Participants; unit: Participants]
  Toxin Naive | 39
  Non-toxin Naive | 81

OUTCOME MEASURES:

1. Primary Outcome: Subject Satisfaction When Treated With abobutulinumtoxinA in Their Glabellar Lines
Description: Percentage of subjects satisfied with the treatment results assessed by satisfaction question at Month 12 visit.
Time Frame: 12 months
Population: Modified Intent to Treat Population (all subjects treated with study product both at Baseline and Month 6) attending Month 12 visit.
Measure: Count of Participants; unit: Participants
Arm/Group | AbobotulinumtoxinA
Number analyzed (Participants) | 110
Participants
  Highly satisfied | 66
  Satisfied | 38
  Dissatisfied | 4
  Highly dissatisfied | 2

2. Secondary Outcome: Subject Satisfaction With Aesthetic Outcome in Treated Area
Description: based on Subject Satisfaction questionnaire data
Time Frame: Months 1,3,6,7,9 and 12
Population: Intent to Treat population (all subjects treated with study product). Number analyzed = Number of subjects completing Subject Satisfaction questionnaire at each visit following treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | AbobotulinumtoxinA
Number analyzed (Participants) | 117
Participants
  Month 1: Very satisfied | 83
  Month 1: Satisfied | 32
  Month 1: Dissatisfied | 2
  Month 1: Very dissatisfied | 0
  Month 3: number analyzed (Participants) | 115
  Month 3: Very satisfied | 44
  Month 3: Satisfied | 55
  Month 3: Dissatisfied | 14
  Month 3: Very dissatisfied | 2
  Month 6: number analyzed (Participants) | 113
  Month 6: Very satisfied | 35
  Month 6: Satisfied | 50
  Month 6: Dissatisfied | 23
  Month 6: Very dissatisfied | 5
  Month 7: number analyzed (Participants) | 106
  Month 7: Very satisfied | 78
  Month 7: Satisfied | 26
  Month 7: Dissatisfied | 2
  Month 7: Very dissatisfied | 0
  Month 9: number analyzed (Participants) | 111
  Month 9: Very satisfied | 61
  Month 9: Satisfied | 40
  Month 9: Dissatisfied | 8
  Month 9: Very dissatisfied | 2
  Month 12: number analyzed (Participants) | 110
  Month 12: Very satisfied | 43
  Month 12: Satisfied | 49
  Month 12: Dissatisfied | 16
  Month 12: Very dissatisfied | 2

3. Secondary Outcome: Evaluate Subject Satisfaction; Appraisal of Lines - Between Eyebrows
Description: FACE-Q Appraisal of Lines: Between Eyebrows. Scored questionnaire to assess treatment outcome from subject's perspective. Minimum Rasch-transformed score = 0; Maximum Rasch-transformed score = 100. Higher score = better outcome.
Time Frame: Months 1,3,6,7,9 and 12
Population: Intent to Treat Population (all subjects treated with study product) attending visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | abobotulinumtoxinA
Number analyzed (Participants) | 120
score on a scale
  Baseline | 31.6 (18.22)
  Month 1: number analyzed (Participants) | 117
  Month 1 | 83.3 (19.22)
  Month 3: number analyzed (Participants) | 115
  Month 3 | 64.2 (22.46)
  Month 6: number analyzed (Participants) | 113
  Month 6 | 44.7 (20.78)
  Month 7: number analyzed (Participants) | 106
  Month 7 | 85.5 (17.77)
  Month 9: number analyzed (Participants) | 111
  Month 9 | 70.7 (23.23)
  Month 12: number analyzed (Participants) | 110
  Month 12 | 51.5 (22.18)

4. Secondary Outcome: Evaluate the Impact of Treatment; Psychological Function
Description: FACE-Q Psychological Function. Scored questionnaire to assess treatment outcome from subject's perspective. Minimum Rasch-transformed score = 0; Maximum Rasch-transformed score = 100. Higher score = better outcome.
Time Frame: Months 1,3,6,7,9 and 12
Population: Intent to Treat Population (all subjects treated with study product) attending visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | abobotulinumtoxinA
Number analyzed (Participants) | 120
score on a scale
  Baseline | 72.2 (22.56)
  Month 1: number analyzed (Participants) | 117
  Month 1 | 84.0 (15.94)
  Month 3: number analyzed (Participants) | 115
  Month 3 | 81.6 (17.29)
  Month 6: number analyzed (Participants) | 113
  Month 6 | 78.0 (20.35)
  Month 7: number analyzed (Participants) | 106
  Month 7 | 85.1 (17.60)
  Month 9: number analyzed (Participants) | 111
  Month 9 | 82.7 (19.02)
  Month 12: number analyzed (Participants) | 110
  Month 12 | 79.0 (17.46)

5. Secondary Outcome: Subject Self-Assessment Using a 4-point Categorical Scale
Description: Evaluate efficacy using a subject self-assessment scale that measures the severity of glabellar lines at maximum frown
Time Frame: Months 1,3,6,7,9 and 12
Population: Intent to Treat Population (all subjects treated with study product) attending visit.
Measure: Count of Participants; unit: Participants
Arm/Group | abobotulinumtoxinA
Number analyzed (Participants) | 120
Participants
  Baseline: Severe | 78
  Baseline: Moderate | 42
  Baseline: Mild | 0
  Baseline: None | 0
  Month 1: number analyzed (Participants) | 117
  Month 1: Severe | 0
  Month 1: Moderate | 10
  Month 1: Mild | 54
  Month 1: None | 53
  Month 3: number analyzed (Participants) | 115
  Month 3: Severe | 12
  Month 3: Moderate | 50
  Month 3: Mild | 45
  Month 3: None | 8
  Month 6: number analyzed (Participants) | 113
  Month 6: Severe | 55
  Month 6: Moderate | 48
  Month 6: Mild | 10
  Month 6: None | 0
  Month 7: number analyzed (Participants) | 106
  Month 7: Severe | 0
  Month 7: Moderate | 14
  Month 7: Mild | 36
  Month 7: None | 56
  Month 9: number analyzed (Participants) | 111
  Month 9: Severe | 9
  Month 9: Moderate | 31
  Month 9: Mild | 53
  Month 9: None | 18
  Month 12: number analyzed (Participants) | 110
  Month 12: Severe | 34
  Month 12: Moderate | 57
  Month 12: Mild | 19
  Month 12: None | 0

6. Secondary Outcome: Investigator Live Assessment Using a 4-point Photographic Scale of Glabellar Line Severity
Description: Evaluate efficacy at visits using a 4-point photographic scale of glabellar line severity, by Investigator Live assessment at maximum frown.
Time Frame: Months 1,3,6,7,9 and 12
Population: Intent to Treat Population (all subjects treated with study product) attending visit.
Measure: Count of Participants; unit: Participants
Arm/Group | abobotulinumtoxinA
Number analyzed (Participants) | 120
Participants
  Baseline: Severe | 82
  Baseline: Moderate | 38
  Baseline: Mild | 0
  Baseline: None | 0
  Month 1: number analyzed (Participants) | 117
  Month 1: Severe | 0
  Month 1: Moderate | 2
  Month 1: Mild | 24
  Month 1: None | 91
  Month 3: number analyzed (Participants) | 115
  Month 3: Severe | 8
  Month 3: Moderate | 27
  Month 3: Mild | 57
  Month 3: None | 23
  Month 6: number analyzed (Participants) | 113
  Month 6: Severe | 50
  Month 6: Moderate | 47
  Month 6: Mild | 16
  Month 6: None | 0
  Month 7: number analyzed (Participants) | 106
  Month 7: Severe | 0
  Month 7: Moderate | 3
  Month 7: Mild | 22
  Month 7: None | 81
  Month 9: number analyzed (Participants) | 111
  Month 9: Severe | 2
  Month 9: Moderate | 30
  Month 9: Mild | 45
  Month 9: None | 34
  Month 12: number analyzed (Participants) | 110
  Month 12: Severe | 35
  Month 12: Moderate | 57
  Month 12: Mild | 16
  Month 12: None | 2

7. Secondary Outcome: Onset of Treatment Response
Description: Subject perception of treatment response
Time Frame: After treatment at Baseline and Month 6, assessed up to 1 week after each treatment visit
Population: Intent to Treat Population (all subjects treated with study product) who returned diary cards.
Measure: Mean (Standard Error); unit: days
Arm/Group | abobotulinumtoxinA
Number analyzed (Participants) | 116
days
  Following Baseline Treatment | 2.5 (0.14)
  Following Month 6 Treatment: number analyzed (Participants) | 107
  Following Month 6 Treatment | 2.4 (0.12)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | AbobotulinumtoxinA
All-Cause Mortality (participants affected / at risk) | 0/120
Serious Adverse Events (participants affected / at risk) | 2/120
Other Adverse Events (participants affected / at risk) | 0/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AbobotulinumtoxinA (N=120)
Abdominoplasty (Surgical and medical procedures) | 1 (1) — hospitalization following abdominoplasty surgery Unrelated to study product or injection procedure Moderate in intensity
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 (1) — Hospitalization for bleeding following abdominoplasty surgery Unrelated to study product or injection procedure Severe in intensity
Ureterolithiasis (Renal and urinary disorders) | 1 (1) — Unrelated to study product or injection procedure Moderate in intensity

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs agree not to present or publish any data or reports collected individually or by subgroup of sites prior to full, initial publication based on all data obtained from all sites.

DOCUMENTS (2):
  • Study Protocol (2018-08-03): https://cdn.clinicaltrials.gov/large-docs/36/NCT03687736/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-04): https://cdn.clinicaltrials.gov/large-docs/36/NCT03687736/SAP_001.pdf